CLINICAL TRIAL: NCT05018117
Title: Effects of Nicotine and Attention on Frequency Tuning in Auditory Cortex
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2018-12-11682; R01AG067073-01A1 (NIH)
Record Dates: First submitted 2021-08-11; First posted 2021-08-24 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Aging
Keywords: nicotine; acetylcholine; functional magnetic resonance imaging
MeSH Terms: interventions — Nicotine Chewing Gum; Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Nicotine (6 mg, polacrilex gum) and placebo will be administered to each participant in separate sessions in a within-subject double-blind randomized crossover design. Subjects will be in either a young (18-28 years) or old (60-85 years) group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Young (18-28 years) participants - nicotine gum (Experimental): 6 mg nicotine gum, one time before fMRI measurements
  Interventions: Drug: Nicotine gum
- Old (60-85 years) participants - nicotine gum (Experimental): 6 mg nicotine gum, one time before fMRI measurements
  Interventions: Drug: Nicotine gum
- Young (18-28 years) participants - placebo gum (Placebo Comparator): placebo gum, one time before fMRI measurements
  Interventions: Other: Placebo gum
- Old (60-85 years) participants - placebo gum (Placebo Comparator): placebo gum, one time before fMRI measurements
  Interventions: Other: Placebo gum

INTERVENTIONS:
Drug: Nicotine gum — The effects of over-the-counter nicotine gum will be compared to a placebo gum
  Other Names: polacrilex
  Arms: Old (60-85 years) participants - nicotine gum; Young (18-28 years) participants - nicotine gum
Other: Placebo gum — The effects of over-the-counter nicotine gum will be compared to a placebo gum
  Arms: Old (60-85 years) participants - placebo gum; Young (18-28 years) participants - placebo gum

SUMMARY:
Nicotine enhances auditory-cognitive function because it mimics the brain's system for "paying attention" to important sounds amid distractions (for example, understanding speech in a noisy environment). In part, nicotine does this by activating inhibitory neurons in the auditory cortex. Since age-related hearing deficits result, in part, from the loss of inhibitory neurons in auditory cortex, this project will determine whether nicotine's effects can compensate for reduced inhibition in the aging auditory cortex and thereby restore auditory function.

The investigators will use functional magnetic resonance imaging (fMRI) to measure the selectivity of responses in auditory cortex to tones of various frequencies. The investigators will measure the effects of nicotine (administered as chewing gum) and aging on these fMRI response properties. The investigators hypothesize that frequency selectivity will decrease with aging and increase following nicotine administration.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers with a score of 0-2 out of 10 maximum on the Fagerström index of smoking dependency

Exclusion Criteria:

* deafness or excessive hearing loss
* smokers with a score between 3 and 10 on the Fagerström index of smoking dependency
* history of psychiatric illness, neurological disorders, diabetes mellitus, renal failure, or cardiovascular disease
* regular use of prescription medications (excluding oral contraceptives)
* drug dependency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
frequency tuning of excitatory auditory fMRI cortical responses | Functional MRI recordings will begin approximately 30 minutes after oral administration of polacrilex or placebo gum and will continue for up to two hours.
  Functional magnetic resonance imaging (fMRI) responses to pure tone stimuli ranging from 88-8000 Hz will be recorded. For each voxel in objectively identified auditory cortical area, a tuning curve model will be fit to the data. One of the parameters of this model is the width of frequency tuning of excitatory responses, and this is the primary outcome measure.

SECONDARY OUTCOMES:
frequency tuning of inhibitory auditory fMRI cortical responses | Functional MRI recordings will begin approximately 30 minutes after oral administration of polacrilex or placebo gum and will continue for up to two hours.
  Functional magnetic resonance imaging (fMRI) responses to pure tone stimuli ranging from 88-8000 Hz will be recorded. For each voxel in objectively identified auditory cortical area, a tuning curve model will be fit to the data. One of the parameters of this model is the width of frequency tuning of inhibitory responses, and this is Outcome 2.
amplitude of excitatory auditory fMRI cortical responses | Functional MRI recordings will begin approximately 30 minutes after oral administration of polacrilex or placebo gum and will continue for up to two hours.
  Functional magnetic resonance imaging (fMRI) responses to pure tone stimuli ranging from 88-8000 Hz will be recorded. For each voxel in objectively identified auditory cortical area, a tuning curve model will be fit to the data. One of the parameters of this model is the amplitude of excitatory responses, and this is Outcome 3.
amplitude of inhibitory auditory fMRI cortical responses | Functional MRI recordings will begin approximately 30 minutes after oral administration of polacrilex or placebo gum and will continue for up to two hours.
  Functional magnetic resonance imaging (fMRI) responses to pure tone stimuli ranging from 88-8000 Hz will be recorded. For each voxel in objectively identified auditory cortical area, a tuning curve model will be fit to the data. One of the parameters of this model is the amplitude of inhibitory responses, and this is Outcome 4.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Silver, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No